CLINICAL TRIAL: NCT07351149
Title: An International Multicentre Prospective Study of Postoperative Acute Kidney Injury in Hospitalized Paediatric Patients
Brief Title: Postoperative Acute Kidney Injury in Children Undergoing Major Non-cardiac Surgery
Acronym: POAKIDS
Status: Not yet recruiting | Type: Observational
Sponsor: Uppsala University (Other)
Collaborators: Uppsala University Hospital (Other); Karolinska Institutet (Other); Skane University Hospital (Other); Karolinska University Hospital (Other); Istituto Giannina Gaslini (Other); Queen Silvia Children's Hospital, Gothenburg, Sweden (Other); Feculdade de Medicina da Universidade de Sao Paulo - Brasil (Other); University of Belgrade (Other); University Hospital, Basel, Switzerland (Other); Hospices Civils de Lyon (Other); University of Bern (Other); University Hospital, Geneva (Other); Royal Perth Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: POAKIDS-2025-04168-02
Record Dates: First submitted 2026-01-09; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-12

CONDITIONS: Acute Kidney Injury
Keywords: Postoperative acute kidney injury; Pediatric kidney injury; Pediatric renal failure; Urinary biomarkers; Pediatric urinary biomarkers; Pediatric postoperative kidney injury; Pediatric anesthesia; Risk factors for pediatric acute kidney injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Urine Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children undergoing major non-cardiac surgery under general anaesthesia: Eligible participants are children aged 0-16 years admitted for non-ambulatory, non-cardiac major surgery requiring general anaesthesia with an estimated duration of at least 60 minutes, including elective, urgent, and emergency procedures. Non-ambulatory surgery is defined as a planned overnight hospital admission following the procedure.

SUMMARY:
This project aims to conduct an international, prospective, multicentre, observational study to determine the incidence of Postoperative Acute Kidney Injury (PO-AKI) in hospitalized children after noncardiac surgery. Urinary biomarkers are intended to be evaluated as predictors of PO-AKI in the same subjects. The study employs modern standardized classifications for AKI to comprehensively address the issue of PO-AKI in children. Describing the incidence and identifying risk factors for PO-AKI will play a crucial role in developing preventive strategies aimed at reducing associated mortality and morbidity. Furthermore, investigating the relationship between urinary biomarkers of renal injury and PO-AKI will provide valuable insights into assessing postoperative renal function in paediatric patients, especially when repeated blood sampling is not feasible.

DETAILED DESCRIPTION:
INTRODUCTION Acute Kidney Injury refers to a sudden impairment in renal function, reflected by increased plasma creatinine concentration and/or decreased urine output. Traditionally, only the most severe reduction in renal function with azotemia and anuria has been emphasised as significantly deleterious, but during the last decades evidence suggests that acute, relatively mild or moderate injury to the kidney portend serious clinical consequences. In critical illness, AKI is strongly associated with short-term mortality as well as chronic kidney disease, cardiovascular disease, and premature death, even when kidney function has recovered.

PO-AKI is characterized by a sudden and significant decline in renal function after surgery. In adults, it is established that PO-AKI is common, imposes a heavy burden of illness, is amenable to early detection and potential prevention and infers a high cost per person in management. There is also considerable variability in practice to prevent, diagnose, treat and achieve outcomes of AKI [1]. Detailed knowledge of incidence rates, risk factors, and outcomes of PO-AKI have considerably enhanced our understanding of optimal treatment and prevention strategies.

Compared to the adult population, there remains a paucity of research data pertaining to PO-AKI for noncardiac surgery in children. However, there is a rational presumption that identifying, preventing, and treating a condition like PO-AKI, which carries enduring long-term consequences, would be particularly advantageous in paediatric patients. The known high burden of AKI in children who are critically ill or undergoing cardiac surgery underscore the importance of accurately and prospectively describing incidence and risk factors for paediatric PO-AKI.

Contemporary evidence advocates for the utilization of innovative urinary biomarkers in predicting and managing AKI. Nevertheless, additional studies are imperative to advance scientific and clinical comprehension regarding the optimal methods and timing for their application, not the least in the perioperative setting. The clinical promise of these biomarkers is particularly pronounced in paediatric populations due to the considerable impediment posed by the necessity for frequent blood sampling in diagnosing and staging PO-AKI within this group. Further investigation stands to enhance the understanding and implementation of these biomarkers, offering substantial potential benefits in the management of paediatric PO-AKI. However, data regarding PO-AKI in paediatric patients, especially those undergoing noncardiac surgery, are notably limited.

RESEARCH QUESTIONS

1. What is the incidence of paediatric PO-AKI in hospitalized children after noncardiac surgery?
2. Can urinary biomarkers, novel and established, accurately predict paediatric PO-AKI?
3. What are the risk factors for AKI in children undergoing anaesthesia and surgery?

THE NEED FOR THE RESEARCH In adults, the impact of PO-AKI is extensively documented. Research indicates a notable disparity in the incidence of kidney failure among individuals who experience PO-AKI compared to those who do not. Specifically, at the one-year mark, the occurrence of kidney failure stands at 0.94% in individuals who have encountered PO-AKI, as opposed to a significantly lower rate of 0.05% in those without such a history. This trend persists over a decade, with kidney failure presenting in 0.4% of patients devoid of renal impairment post-surgery, whereas 2.3% of those affected by PO-AKI develop kidney failure within the same period. PO-AKI also further impair an already reduced renal function. While 7.3% of patients with Chronic Kidney Disease (CKD) progress to kidney failure over ten years, this figure elevates to 15.7% for individuals with CKD who have experienced PO-AKI. Even when kidney function fully recovers, individuals with a history of PO-AKI exhibit persistently inferior survival rates over a ten-year period. Additionally, patients who undergo PO-AKI face heightened risks of recurrent AKI episodes and future reliance on renal replacement therapy. Various postoperative complications, such as infections, prolonged mechanical ventilation, tracheostomy, and cardiovascular events, are more prevalent among patients who develop PO-AKI post-surgery compared to those who do not. Furthermore, PO-AKI incurs substantial hospitalization costs and increased utilization of resources. Thus, in adults PO-AKI pose a serious problem.

PAEDIATRIC POSTOPERATIVE ACUTE KIDNEY INJURY Millions of children undergo various surgical procedures globally each year, ranging from routine to complex surgeries. Limited research has focused on paediatric PO-AKI using contemporary criteria for renal dysfunction in noncardiac surgery. The majority of existing studies are retrospective, single-centre investigations reporting widely varied incidence of PO-AKI, ranging from 3.2% to 62.3%. Only one study is from Europe and two are prospective. Importantly, several studies focus solely on neonatal PO-AKI.

Large, well-performed studies in critically ill neonates and children demonstrate an incidence of AKI at rates of 29% and 27%, respectively. After paediatric cardiac surgery AKI is also common, although the prevalence is highly variable among different investigations. The estimated incidence is somewhere between 15%-60%, although a recent single-centre study using the KDIGO-criteria presented an incidence of 9.3%. AKI in neonates and children, regardless of triggering event, significantly correlates with in-hospital mortality and prolonged hospital stays. The long-term consequences of renal failure have been described as hypertension, proteinuria and chronic kidney disease, which is alarming since chronic renal pathology in youth is known to have extensive adverse effects.

URINARY BIOMARKERS OF RENAL DAMAGE Current diagnosis and staging of AKI rely on changes in plasma creatinine concentration or urine output. However, using plasma creatinine as a biomarker for renal dysfunction in the paediatric population presents several challenges. In early life, plasma creatinine levels primarily reflect maternal levels and are expected to decrease during the initial postnatal week. A failure of creatinine levels to decrease might signify impaired renal function, which may not be identified using the KDIGO definition. Additionally, plasma creatinine is a delayed marker of kidney function and may not accurately reflect minor renal impairment. Blood sampling, a requirement for diagnosis, poses practical and ethical challenges in children. These impediments collectively contribute to the problems in defining the incidence of PO-AKI and developing successful clinical trials and interventions for paediatric AKI.

Novel urinary biomarkers initially identified in high-risk populations show promise in early and precise diagnosis of paediatric AKI, potentially surpassing plasma creatinine analysis. However, there remains a lack of studies validating their use. A recent consensus statement recommends employing a combination of damage and functional biomarkers, along with clinical information, to identify high-risk patient groups, enhance AKI diagnosis, optimize care processes, and aid AKI management. Nevertheless, the same consensus statement also acknowledges that substantial knowledge gaps persist, necessitating further research. One significant obstacle in using urinary biomarkers for AKI is the release of endogenous substances during inflammation, clouding the interpretation of biomarker concentration increases in immune-stimulated patients. However, these challenges may be less significant in PO-AKI as children generally have fewer comorbidities and thus less acute/ chronic inflammation. Additionally, the timing of potential renal insults (anaesthesia and surgery) is known and can be accounted for. Different biomarkers reflecting increased urinary concentrations indicate damage at various nephron levels (See Fig 2). Thus, if properly evaluated urinary biomarkers may prove to be an accurate and useful predictor of PO-AKI and also give mechanistic insight into the cause of the renal injury.

RISK FACTORS OF PAEDIATRIC POSTOPERATIVE ACUTE KIDNEY INJURY Several risk factors contribute to paediatric PO-AKI beyond the inflammatory response induced by surgery per se. Events in the perioperative setting, such as hypotension, hypoxia, infections, mechanical ventilation, fluid shifts, blood loss and exposure to nephrotoxic medications, are potential culprits. Renal hypoperfusion due to hypotension may occur due to various reasons, including hypovolemia due to blood loss or dehydration after fasting and inflammation-induced capillary leak. In adults it has been demonstrated that intraoperative hypotension is associated with AKI in noncardiac surgical populations. Longer hypotensive periods and lower blood pressure results in higher AKI probabilities. Infants with vasopressor treatment or high fluid infusion rates during abdominal surgery have higher risk of AKI compared with those without blood pressure support [22]. Another potential risk factor is the choice of anaesthetic. It was demonstrated that volatile anaesthesia, compared with total intravenous propofol anaesthesia, is associated with reduced urine output and higher incidence of PO-AKI in adults. Finally, it was recently described that female sex confers protection against AKI. This has not previously been examined in a paediatric population or in the perioperative setting.

ELIGIBILITY:
Inclusion Criteria:

* Elective, urgent or emergency in-patient major non-cardiac surgical procedures performed under general anaesthesia with or without regional analgesia with a planned procedure duration of at least 60 minutes.
* Paediatric patients (0-16 years old)

Exclusion Criteria:

* Declined participation.
* Ongoing renal replacement therapy
* Acute Kidney Injury (according to KDIGO)
* Known chronic kidney disease
* Procedure involving surgery of the kidney
* Procedures requiring clamping of blood flow to or from the kidney
* Body weight <2kg
* Procedure involving contrast administration
* Established rhabdomyolysis (CK-levels >1500 U/L)

Ages: 0 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Hospitalised paediatric patients undergoing major non-cardiac surgery in any of the specified investigator sites
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of postoperative AKI | Within 7 postoperative days
  Incidence of postoperative AKI, defined according to the Kidney Disease: Improving Global Outcomes (KDIGO) creatinine criteria, based on changes in plasma/serum creatinine concentration from baseline within the postoperative period:
  * AKI Stage 1: Increase in plasma/serum creatinine ≥ 0.3 mg/dL (26.5 µmol/L) within 48 hours postoperatively OR 1.5-1.9 times baseline plasma/serum creatinine within 7 postoperative days.
  * AKI Stage 2: Increase in plasma/serum creatinine 2-2.9 times baseline p/s creatinine within 7 postoperative days.
  * AKI Stage 3: Increase in plasma/serum creatinine > 3 times baseline plasma/serum creatinine within 7 postoperative days OR increase in plasma/serum creatinine to 4.0mg/dL (353.6 µmol/L) OR Initiation of renal replacement therapy OR decrease in eGFR to < 35mL/min per 1.73 m2. All within 7 postoperative days.
  Baseline creatinine is defined as a plasma/serum creatinine value obtained within 24 hours prior of commencement of surgery.

SECONDARY OUTCOMES:
Agreement and association between changes in plasma/serum creatinine and urinary biomarkers of renal injury. | Within 7 postoperative days
Time from surgery to first AKI-qualifying creatinine | Within 7 postoperative days
Perioperative risk factors associated with postoperative AKI | Within 7 postoperative days
Diagnostic accuracy of plasma cystatin C for postoperative AKI and agreement with creatinine-based definitions. | Within 7 postopertive days
Associations between AKI and mortality, length of stay and renal replacement therapy | Within 7 postoperative days

OTHER OUTCOMES:
Incidence of postoperative dysnatraemia and associated risk factors | Within 7 postoperative days
Incidence of postoperative dyschloremia and associated risk factors. | Within 7 postoperative days
Incidence of postoperative dyskalemia and associated risk factors. | Within 7 postoperative days
Incidence of postoperative AKI defined by urine output | Within 3 postoperative days
  Urine output criteria for AKI will be recorded where available, but creatinine-based KDIGO criteria constitute the primary diagnostic definition.
  o If patient age at time of surgery ≥ 28 days: AKI Stage 1: <0.5 mL/kg/h for 6-12h AKI Stage 2: <0.5 mL/kg/h for ≥ 12h AKI Stage 3: <0.3 mL/kg/h for ≥24h or anuria ≥12h
  o If patient age at time of surgery < 28 days: AKI Stage 1: <1 mL/kg/h for ≥24h AKI Stage 2: <0.5 mL/kg/h for ≥24h AKI Stage 3: <0.3 mL/kg/h for ≥24h or anuria ≥12h

CONTACTS AND LOCATIONS:
Overall Officials: Robert Frithiof, MD, PhD, Principal Investigator — Uppsala University Hospital, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data underlying the results reported in publications from the POAKIDS study, including baseline characteristics, perioperative variables, outcome data, and biomarker measurements. All data will be fully anonymised at the individual level so that no participant can be identified.
Supporting Information: Study Protocol
Time Frame: Data will be available beginning 12 months after publication of the primary results and will remain available upon reasonable request for at least 5 years thereafter.
Access Criteria: Access to the de-identified dataset will be granted to qualified researchers upon reasonable request. Requests must include a brief description of the research question, analysis plan, and intended use of the data. All requests will be reviewed by the POAKIDS steering committee. Data will be shared only for scientifically sound projects and for purposes consistent with the original study objectives and ethical approvals. Data will be shared through secure data transfer following approval of a data sharing agreement. No direct identifiers or site-specific identifiers will be included in the shared dataset.

REFERENCES:
- See also: Related Info — https://www.uu.se/poakids